CLINICAL TRIAL: NCT01490138
Title: Investigation of the Clinical Relevance of Serial Concentrations of β-D-Glucan Tests in the Patients With Invasive Fungal Infection
Brief Title: Investigation of Clinical Relevance of β-D-Glucan Tests in Patients With Invasive Fungal Infection (IFI)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ruijin Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Other Study IDs: G-test and IFI
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Fungal Infection
Keywords: β-D-Glucan test; IFI
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Invasive fungal infection (IFI) is a disease usually occurred in the patients with compromised immune condition, such as acute leukemia, allogeneic stem cell transplantation or long term immune suppression treatment with the incidence increasing over last decades. Given the introduction of numerous anti-fungal agents and great advance has been made in recent years, IFI is still a dangerous disease with high mortality.

Early diagnosis of IFI is still a problem challenging the physicians. Serum tests of β-D-Glucan are introduced to the diagnosis of IFI, which have the advantage of easy application. However, the value of this test in the monitoring of antifungal treatment remains unclear.

The investigators perform this study to evaluate the correlation of the serum test results of β-D-Glucan test with the treatment response during the anti-fungal treatment, and hope to see that the results of serial serum tests are good predictive markers for treatment response.

DETAILED DESCRIPTION:
This is a single center, open-label study. The duration of the study will be 2 years. The number of targeted subjects will be 50 (in 2 years). We estimate that on average, the treatment duration is 4-8 weeks. Serum Glucan levels will be measured 2 times per week until the recovery of the infection or treatment end.

ELIGIBILITY:
Inclusion Criteria:

Patients with proven or probable IFI and immunocompromised because of hematopoietic-cell transplantation (HSCT) or chemotherapy, and have positive results for serum Glucan tests will be included in the study.

Patients must satisfy all the following criteria before entering the study :

1. Episode of proven or probable IFI, diagnosed according to the EORTC/MSG definitions;
2. Immunocompromised because of HSCT or chemotherapy for malignant hematopathy;
3. ≥ 2 consecutive positive serum glucan level, using a threshold for positivity of ≥ 60 ng/L, at the start of antifungal therapy.

Exclusion Criteria:

If the fungal infection of the patient is excluded or confirmed to be a specific pathogen other than fungi before the enrollment/during the study period, he or she will be excluded/withdrew from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with compromised immune condition, such as acute leukemia, lymphoma, myeloma, allogeneic stem cell transplantation or long term immune suppression treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Weili ZHAO, PhD, Principal Investigator — Ruijin Hospital